CLINICAL TRIAL: NCT03367208
Title: Study of Metabolites Markers in Adjuvant Breast Cancer
Acronym: EMMEEA
Status: Completed | Type: Observational
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/07
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2017-12

CONDITIONS: Breast Neoplasms
Keywords: metabolomic
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: frozen surgery specimen, frozen serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The breast cancer is composed of multiple biological entities. Recent progress in molecular biology, DNA or RNA chip, permitted the global tumour genome or transcriptome study. Those technics, leads to an increased in the molecular biology knowledge and a better oncogenesis understanding. Breast cancer taxonomy was established following the tumor genetic profile. Moreover this classification is incomplete and didn't include the metabolic pathways other than hormonal or HER2 pathways.

The metabolomics is an expanding field of research exploring the metabolites in cells, tissues or biologics fluids. It allows assessing the variation activation of the different cellular metabolic pathways. In oncology, it could highlight the main metabolic disturbances, the interaction of tumor cells and to identify the metabolic pathways involved in oncogenesis using the tumor cells metabolites profiles.

Compared to genomic, the metabolomics integrated the impact of the cells environments on the cells biology. The cells environment plays, in fact, a key role in the oncogenesis and in the tumor cells phenotypes. The metabolomics, thus being a complementary approach of the genomic in order to assess a better knowledge of the impact of the extracellular environment on the tumor cell phenotype. In addition, the metabolomics analyses are fast and not expensive compatible with routine practice.

The main objective of this study is to highlight a metabolic alteration specific to certain tumors phenotypes in order to have better understanding of the biology of the numerous breast cancer entities and find some biomarkers which could be some possible therapeutic target. Using a high resolution mass spectrometer, the investigators will analyze 52 tumor samples from frozen breast surgical specimen preserved in the Centre Antoine lacassagne tumor bank. The tissue analysis could be associated with a serum sample analysis from the frozen serum bank of the Centre Antoine Lacassagne. With 30 patients who performed a 18 FDG-PET before the surgery, The investigators will analyzed the correlation between the tumoral activation of the glycolysis pathways, quantified with mass spectroscopy and the 18FDG uptake. Using the 17 frozen serums available, the investigators will perform a screening to identify some metabolites or metabolites profile which could be detected in the serum in order to develop a new liquid biopsy approach. This study is a retrospective study based on data and sample already available in the center and collected during the routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Patient with breast cancer who undergoes a initial surgery with frozen preservation of the surgical specimen in the Centre Antoine Lacassagne tumor bank
* Patient who sign the Biological research center consent allowing the the preservation of tumor and blood sample in biobank and use of the sample for research purpose

Exclusion Criteria:

* other treatment the initial surgery (neodjuvant chemotherapy...)
* Absence of tumor tissue available in the tumor bank
* Absence of Biological research center consent signed

Min Age: 10 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who undergoes a initial surgery for a breast cancer in the Centre Antoine Lacassagne with surgical specimen available for the research
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Metabolomic profil diagnosis value | april 2017

SECONDARY OUTCOMES:
correlation coefficient between glycolysis pathway metabolic concentration and 18FDG uptake | april 2017
qualitative profile of tumor metabolic in serum | april 2017
quantitative profile of tumor metabolic in serum | april 2017
PFS comparisons at 2 years regarding the presence or absence of some metabolites (serum or tissue) | 2 years
Test of concordance between metabolites found in tissues and serum sample | april 2017

CONTACTS AND LOCATIONS:
Overall Officials: Christine LOVERA, Study Director — Centre Anointe Lacassagne
Locations (1):
- Centre Antoine Lacassagne, Nice, Cedex 2, France